CLINICAL TRIAL: NCT06991400
Title: Evaluation of Laparotomy With Trans-Amniotic Suture Placement in TTTS Surgery
Acronym: TTTS TAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Foong-Yen Lim, Surgical Director, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0006
Record Dates: First submitted 2024-11-02; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Twin to Twin Transfusion Syndrome; Twin Anemia-Polycythemia Sequence
Keywords: fetoscopic surgery, laparotomy
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- yes stitch (will receive a larger stitch from laparotomy) (Experimental): yes stitch for a larger stitch when receiving a laparotomy.
  Interventions: Other: Trans-Amniotic Suture Placement
- No stitch (No Intervention)

INTERVENTIONS:
Other: Trans-Amniotic Suture Placement — Trans-Amniotic Suture placement
  Arms: yes stitch (will receive a larger stitch from laparotomy)

SUMMARY:
This is a randomized trial for patients that are diagnosed with Twin-Twin Transfusion Syndrome (TTTS) who are receiving a fetoscopic laser surgery to evaluate the effectiveness and safety of a laparotomy closure.

DETAILED DESCRIPTION:
The rationale behind suturing the hole is that the amniotic membrane does not close itself, rather you are relying that the uterus closes over the hole in the amniotic membrane, which may or may not happen, as well as in fetoscopic surgery for another condition, myelomeningocele. Published data has shown that maternal laparotomy to suture closure of the port site at the time of fetoscopic surgery leads to improved pregnancy outcomes, later gestational age at delivery, and lower rates of preterm pre-labor rupture of membranes (PPROM) [PMID: 28910784].

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of TTTS or Twin Anemia-Polycythemia Sequence (TAPS)
* Gestational age between 18 weeks and 23 weeks (18 0/7 to 22 6/7 weeks)
* Cervical length >2.5 cm preoperatively
* Identification of a safe percutaneous surgical window by a provider experienced in fetoscopic surgery prior to entering the operating room

Exclusion Criteria:

* Higher order pregnancies, chromosomal or severe congenital anomalies, undergoing laser surgery for fetal growth restriction only, need for a second laser during pregnancy, failure to complete laser, PPROM prior to surgery. BMI> 40 at the start of pregnancy, emergent case (i.e. surgery occurs < 6 hours from presentation), significant fetal anomalies expected to drastically alter the risk of neonatal morbidity or mortality (i.e. anencephaly, cyanotic heart disease), or any significant maternal comorbidities as determined by physician i.e.: clotting disorders/blood disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Latency from surgery to delivery | 4 months
  Will a transuterine suture placement cause later gestational age at delivery in babies with TTTs.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We are using the data for CCHMC only.

REFERENCES:
- [Background] Forde B, Sepulveda Gonzalez G, Lim FY, Arroyo-Lemarroy T, Nava Geurrero EN, Lizarraga-Cepeda E, Habli M, McKinney D, Hoffman M, Peiro JL. Should We Stitch-Close the Fetoscopic Percutaneous Access? A Case-Series of Laparotomy to Trans-Amniotic Membrane Suturing for Intrauterine Port Placement in Fetoscopic Surgery for Twins. Fetal Diagn Ther. 2024;51(5):510-515. doi: 10.1159/000539894. Epub 2024 Jun 18. PMID 38889699
- [Background] Kabagambe SK, Jensen GW, Chen YJ, Vanover MA, Farmer DL. Fetal Surgery for Myelomeningocele: A Systematic Review and Meta-Analysis of Outcomes in Fetoscopic versus Open Repair. Fetal Diagn Ther. 2018;43(3):161-174. doi: 10.1159/000479505. Epub 2017 Sep 15. PMID 28910784